CLINICAL TRIAL: NCT01062516
Title: Influence of Esomeprazole on Antiplatelet Action of Clopidogrel Associated With Aspirin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ruttonjee Hospital (Other)
Responsible Party: Dr Fook Hong Ng, Ruttonjee Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: HKEC 2007-176 VerifyNow
Record Dates: First submitted 2010-02-02; First posted 2010-02-04 (Estimated); Last update posted 2010-10-05 (Estimated); Status verified 2010-10

CONDITIONS: Acute Coronary Syndrome; Acute Myocardial Infarction
Keywords: acute coronary syndrome; acute myocardial infarction; percutaneous coronary intervention; aspirin; clopidogrel; esomeprazole; famotidine; platelet function
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Esomeprazole; Famotidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): oral esomeprazole 20 mg daily
  Interventions: Drug: esomeprazole 20 mg daily
- 2 (Active Comparator): oral famotidine 40mg daily
  Interventions: Drug: famotidine 40 mg daily

INTERVENTIONS:
Drug: esomeprazole 20 mg daily — oral famotidine 40 mg daily vs. oral esomeprazole 20 mg daily for 28 days
  Arms: 1
Drug: famotidine 40 mg daily — oral famotidine 40 mg daily vs. oral esomeprazole 20 mg daily for 28 days
  Arms: 2

SUMMARY:
The investigators examine the influence of esomeprazole versus famotidine on antiplatelet action of clopidogrel associated with aspirin. At least 100 consecutive patients suffering from acute coronary syndrome or undergoing coronary artery stent implantation , who received aspirin (80 - 160 mg/day) and clopidogrel (300 mg loading dose, followed by 75 mg/day or 75mg/day for at least 7 consecutive days), are randomised to receive either esomeprazole 20 mg daily vs famotidine 40 mg daily in a double blinded manner. Clopidogrel effect was tested by measuring residual platelet reactivity (RPR) to ADP by VerifyNow P2Y12 assay (Accumetrics Inc, San Diego, Calif). At baseline, whole blood will be obtained for RPR at least 12 h after clopidogrel loading dose or at least 7 days of maintaince dose. Immediately obtaining the baseline blood, patients will be randomized to receive either esomeprazole (20 mg/day) or famotidine 40 mg/day for 28 days. Double blinding will be performed by encapsulation of study drugs. RPR will be measured again at the 28th day.

The investigators will compare the % inhibition and the P2Y12 reaction Units (PRU) at the 28-day treatment period in the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from acute coronary syndrome or undergoing coronary artery stent implantation (PCI) , who received aspirin (80 - 160 mg/day) and clopidogrel (300 mg loading dose, followed by 75 mg/day), are recruited.

Exclusion Criteria:

* known active peptic ulcer disease or gastrointestinal within 8 wk
* known iron deficiency anemia with Hb < 10 gm/dl
* mechanical ventilation
* active cancer, liver cirrhosis, end-stage renal failure
* life expectancy < 1 yr
* known allergic to aspirin, clopidogrel, famotidine or esomeprazole
* pregnancy, lactation, child-bearing potential in the absence of contraception,
* co-prescription of NSAID, corticosteroid, or warfarin
* non-oral feeding or impaired GI absorption e.g. vomiting
* patient on proton pump inhibitor within 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
P2Y12 reaction units | 28 days

SECONDARY OUTCOMES:
percent inhibition | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Fook Hong Ng, MBBS, Principal Investigator — Ruttonjee Hospital
Locations (1):
- Ruttonjee Hospital, Hong Kong, China

REFERENCES:
- [Derived] Tunggal P, Ng FH, Lam KF, Chan FK, Lau YK. Effect of esomeprazole versus famotidine on platelet inhibition by clopidogrel: a double-blind, randomized trial. Am Heart J. 2011 Nov;162(5):870-4. doi: 10.1016/j.ahj.2011.08.007. PMID 22093203